CLINICAL TRIAL: NCT05721235
Title: A Multicenter, Dose-Optimized, Open-Label, Safety/Tolerability and Pharmacokinetic Study With Azstarys® in Children 4 and 5 Years of Age With Attention-Deficit/Hyperactivity Disorder
Brief Title: A Safety/Tolerability and PK Study With Azstarys® in Children With ADHD
Acronym: KP415P02
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Corium, Inc. (Industry)
Collaborators: Premier Research (Other); Prometrika, LLC (Industry); Almac (Industry); Worldwide Clinical Trials (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KP415.P02
Record Dates: First submitted 2023-02-01; First posted 2023-02-09 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Attention Deficit/Hyperactivity Disorder
Keywords: ADHD; Azstarys; Serdexmethylphenidate; Attention Deficit Hyperactvity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Dexmethylphenidate Hydrochloride

STUDY DESIGN:
Intervention Model Description: The primary objective is to determine the safety and tolerability for up to 12 months of treatment with Azstarys based on incidence of adverse events
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open Label (Experimental): 13.1 mg/2.6 mg SDX/d-MPH, 26.1/5.2 mg SDX/d-MPH, or 39.2 mg/7.8 mg SDX/d-MPH
  Interventions: Drug: Serdexmethylphenidate (SDX) and dexmethylphenidate (d-MPH)

INTERVENTIONS:
Drug: Serdexmethylphenidate (SDX) and dexmethylphenidate (d-MPH) — Serdexmethylphenidate (SDX) and dexmethylphenidate (d-MPH)

SUMMARY:
The is a multicenter, dose-optimized, open-label, safety/ tolerability and pharmacokinetic (PK) study with Azstarys® in children 4 and 5 years of age with attention-deficit/hyperactivity disorder (ADHD). The primary objective is to determine the safety and tolerability of treating children 4 and 5 years-of-age with ADHD with Azstarys® for up 12 months. Approximately 100 subjects will be enrolled. Approximately 20 sites will participate.

DETAILED DESCRIPTION:
• Screening Period: New subjects will undergo a Screening Period up to 30 days prior to entering the Dose Optimization Phase.

• Dose Optimization Phase: During the 3-week Dose Optimization Phase, subjects will start at 13.1 mg/2.6 mg, and may be titrated to doses of 26.1 mg/5.2 mg or 39.2 mg/7.8 mg Azstarys® capsules based on individual tolerability and best dose-response in the opinion of the Investigator.

• Treatment Phase: Eligible subjects will receive single daily doses of Azstarys® for approximately 360 ±20 days (approximately 12 months). The starting dose of Azstarys® in the Treatment Phase will be the same as the optimized dose of Azstarys® at the end of the Dose Optimization Phase, either 13.1 mg/2.6 mg, 26.1/5.2 mg, or 39.2 mg/7.8 mg per day. The daily dose may be changed at any time to any of the allowed dose levels (13.1 mg/2.6 mg, 26.1/5.2 mg, or 39.2 mg/7.8 mg per day) at the Investigator' discretion, based on individual tolerability and dose response.

ELIGIBILITY:
Inclusion Criteria:

1. New Subjects must be at least 4 years old and less than 5 years and 10 months old at Screening.
2. Subjects must have a body weight within the 5th and 95th percentile according to the gender-specific weight-for-age percentile charts from the Centers for Disease Control and Prevention (CDC).
3. Subject must be in general good health defined as the absence of any clinically relevant abnormalities as determined by the Investigator based on physical examinations, vital signs, ECGs, medical history, and clinical laboratory values (chemistry, hematology and urinalysis) at Screening.
4. At least one parent/legal guardian of the subject must voluntarily give written permission for the subject to participate in the study.
5. Subject must meet Diagnostic and Statistical Manual of Mental Disorders - Fifth Edition (DSM-5) criteria for a primary diagnosis of ADHD (combined, inattentive, or hyperactive/impulsive presentation) per clinical evaluation and confirmed by the Mini-International Neuropsychiatric Interview for Children and Adolescents (MINI Kid).
6. Subject must have had ADHD symptoms present for at least 6 months prior to the Screening Visit.
7. Subject must be able and willing to wash out current stimulant ADHD medications, including herbal medications from 5 days prior to the start of the Dose Optimization Phase, and abstain from taking these to the end of the Treatment Phase (Visit 17) or Early Termination (ET); and wash out non-stimulant ADHD medications from 14 days prior to the start of the Dose Optimization Phase, and abstain from taking these to the end of the Treatment Phase (Visit 17) or ET.
8. Subject must have a score of ≥4 (Moderately Ill) on the clinician-administered Clinical Global Impressions-Severity (CGI-S) scale.
9. Subject functions at an age-appropriate level intellectually, as determined by the Investigator.
10. Subject must have age and sex adjusted ratings of ≥90th percentile Total Score on the ADHD-RS-IV (Preschool Version) rated over the past 6 months.
11. Subject must have a systolic and diastolic blood pressure below the 95th percentile for age, and gender according to the 2017 AAP guidelines (Flynn 2017) based on the average of 3 measurements 2-5 minutes apart.
12. Subject's parent/legal guardian and caregiver (if applicable) must understand and be willing and able to comply with all study procedures and visit schedule.
13. Subject's parent/legal guardian, and caregiver (if applicable) must be able to speak and understand English or Spanish and be able to communicate satisfactorily with the Investigator and study coordinator.

Exclusion Criteria

1. Subject with any clinically significant chronic medical condition that, in the judgment of the Investigator, may interfere with the participant's ability to participate in the study.
2. Subject has any diagnosis of bipolar I or II disorder, major depressive disorder, conduct disorder, obsessive-compulsive disorder, any history of psychosis, autism spectrum disorder, disruptive mood dysregulation disorder (DMDD), intellectual disability, Tourette's Syndrome, confirmed genetic disorder with cognitive and/or behavioral disturbances.
3. Subject has generalized anxiety disorder or panic disorder that has been the primary focus of treatment at any time during the 12 months prior to Screening, or that has required pharmacotherapy any time during the 6 months prior to Screening.
4. Subject has evidence of any chronic disease of the central nervous system (CNS) such as tumors, inflammation, seizure disorder, vascular disorder, potential CNS related disorders that might occur in childhood (e.g., Duchenne Muscular dystrophy, myasthenia gravis, or other neurologic or serious neuromuscular disorders), or history of persistent neurological symptoms attributable to serious head injury.
5. Subject taking anticonvulsants for seizure control currently or within the past 2 years before Screening are not eligible for study participation.
6. Subject has a current (last month) psychiatric diagnosis other than specific phobia, motor skills disorders, ODD, sleep disorders, elimination disorders, adjustment disorders, learning disorders, or communication disorders.
7. In the opinion of the Investigator, subject has clinically significant suicidal ideation/behavior, based on history of attempted suicide and the C-SSRS assessment at Screening.
8. Subject has any clinically significant unstable medical abnormality, chronic disease (including asthma or diabetes), or a history of a clinically significant abnormality of the cardiovascular (including cardiomyopathy, serious arrhythmias, structural cardiac disorders, or severe hypertension), gastrointestinal, respiratory, hepatic, or renal systems, or a disorder or history of a condition (e.g., malabsorption, gastrointestinal surgery) that may interfere with drug absorption, distribution, metabolism, or excretion of study drug.
9. Subject has a history or presence of abnormal ECGs, which in the Investigator's opinion is clinically significant.
10. Subject has a history of, or currently has a malignancy.
11. Subject has uncontrolled thyroid disorder as evidenced by thyroid stimulating hormone (TSH) ≤0.8 x the lower limit of normal (LLN) or ≥1.25 x the upper limit of normal (ULN) for the reference laboratory at Screening.
12. Subject has greater than trace proteinuria on the urinalysis at Screening.
13. A current or recent (past 12 months) history of drug abuse in someone living in the subjects' home.
14. Subject has a positive urine screen for drugs of abuse at Screening. If the urine test is positive for any of the analytes at Screening, the subject will be excluded from study participation, with the exception of the following: Depending on a subject's current ADHD medication at Screening, the urine screen may test positive for MPH for treatment of their ADHD.
15. Subject has participated in any other clinical study with an investigational drug/product within 30 days or at least 5 half-lives, whichever is longer, prior to Screening, except for participation in Study KP415.P01.
16. Subject has taken ADHD medications from more than one class within 30 days prior to Screening. Subjects on a stable dose of one ADHD medication with occasional use of ADHD medications from another class are eligible at the discretion of the Investigator.
17. Subject has demonstrated lack of response or intolerability to adequate dose and duration of treatment with methylphenidate products.
18. Subject is using or planning to use prohibited drugs during the trial as specified in the protocol.
19. Subject is planning to initiate psychotherapy during the study (subjects participating in psychotherapy beginning at least 4 weeks before study initiation are permitted to continue).
20. Subject has a history of severe allergies or adverse drug reactions to more than one class of medications.
21. Subject has a history of allergic reaction or a known or suspected sensitivity to methylphenidate or any substance that is contained in the study drug.
22. Subject, parent/legal guardian and caregiver (if applicable at the Investigator's discretion) has commitments during the study that would interfere with attending study visits.
23. Subject or subject's family anticipates a move outside the geographic range of the investigative site during the study or plans extended travel inconsistent with the recommended visit interval during study duration.
24. Subject has one or more siblings living in the same household who are enrolled in this or another clinical drug trial.
25. Subject shows evidence of current physical, sexual, or emotional abuse.
26. Subject is, in the opinion of the Investigator, unsuitable in any other way to participate in this study.

Ages: 4 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 123 (Actual)
Dates: Start 2023-06-02 (Actual); Primary Completion 2025-08-29 (Actual); Study Completion 2025-08-29 (Actual)

PRIMARY OUTCOMES:
A determination of safety and tolerability of up to 12 months of treatment with Azstarys | 12 months
  Safety and tolerability will be assessed by the incidence of adverse events reported in the study

CONTACTS AND LOCATIONS:
Overall Officials: Ann Childress, MD, Principal Investigator — Center for Psychiatry And Behavioral Medicine Inc.
Locations (20):
- United States (20):
  - Preferred Research Partners (PRP), Little Rock, Arkansas
  - Advanced Research Center (ARC), Anaheim, California
  - IMMUNOe International Research Center, Centennial, Colorado
  - Clinical Neuroscience Solutions - Orlando, Jacksonville, Florida
  - Accel Research Sites - Lakeland, Lakeland, Florida
  - Accel Research Sites - Maitland, Maitland, Florida
  - South Florida Research Phase I-IV INC, Miami Springs, Florida
  - CNS Healthcare - Orlando, Orlando, Florida
  - iResearch Atlanta, Decatur, Georgia
  - CenExel iResearch, LLC, Savannah, Georgia
  - Sky Clinical Research Network Group P.C., Union City, Georgia
  - DelRicht Research - Touro Medical Center, New Orleans, Louisiana
  - St Charles Psychiatric Associates & Midwest Research Group, Saint Charles, Missouri
  - Boeson Research, Missoula, Montana
  - Alivation Research, LLC, Lincoln, Nebraska
  - Center For Psychiatry and Behavioral Medicine Inc, Las Vegas, Nevada
  - Clinical Neuroscience Solution, Inc, Memphis, Tennessee
  - Houston Clinical Trials, Bellaire, Texas
  - AIM Trials, Plano, Texas
  - Flourish Research, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No